CLINICAL TRIAL: NCT01802450
Title: Multicenter, Open-label, Non-randomized Phase II Trial of Dasatinib in Patients With Chronic Myeloid Leukemia in Chronic Phase (CP-CML) Who Meet Criteria for Late Suboptimal Response After Prior Imatinib Treatment
Brief Title: Dasatinib in Patients With Chronic Myeloid Leukemia in Chronic Phase
Acronym: DASAPOST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PETHEMA Foundation (Other)
Collaborators: Dynamic Solutions (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DASAPOST
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib (Sprycel) (Experimental): Dasatinib (Sprycel): 100 mg QD administered orally as continuous daily dosing (CDD)until disease progression or adverse events that, by protocol definition or Investigator judgment, would preclude further treatment with dasatinib
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib

SUMMARY:
Trial try to assess the efficacy of dasatinib in terms of major molecular response rate at 6 months in patients with CP-CML who have achieved complete cytogenetic response without major molecular response after at least 18 months on Imatinib 400/600.

DETAILED DESCRIPTION:
This is a single-arm, open-label, phase II trial for patients in complete cytogenetic response that have not achieved major molecular response or have lost a prior major molecular response, after at least 18 months of treatment with imatinib.

All enrolled patients will receive dasatinib 100 mg once daily orally for 1 year until progression, loss of cytogenetic response, transformation to advanced phases, unacceptable toxicity (clinical adverse event, lab abnormality or concurrent disease), pregnancy if a female or withdrawal of consent, whichever happens first. Patients will undergo BCR-ABL assessments at study entry and every 3 months (central lab) and immunophenotyping and studies for clonal lymphocytosis at study entry, at 3 and 6 months.

Cytogenetic assessment will be done only if loss of response/progression/clonal evolution are suspected.

Subjects will be evaluated for the efficacy and safety of dasatinib (Sprycel). Lymphocytosis data will be collected for all patients and separate description for efficacy and safety parameters will be done in patients with and without lymphocytosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >or = 18 years
* Diagnostic of Ph+ Chronic Myeloid Leukemia in first chronic phase
* Treated with Imatinib 400 mg per day or 600 mg per day for at least 18 months. A wash out period of at least 7 days for imatinib is required prior to dasatinib administration
* Patients meet criteria of late suboptimal response (complete cytogenetic response with no major molecular response) or have lost major molecular response
* Ability to understand and voluntarily sign the informed consent for
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy and have a negative pregnancy test, a maximum of 72 hours prior to study drug start.

Sexually active men must also use effective contraceptive methods during the treatment.

* Women must not be breastfeeding

Exclusion Criteria:

* Patients treated with Imatinib at a dose different of 400/600 mg per day
* Patients treated with other TKI than imatinib
* Loss of cytogenetic response at study entry
* ECOG ≥ 3
* Inadequate bone marrow reserve: ANC <1.5 x 109/L and/or Platelet count < 100 x 109/L
* Inadequate hepatic function (Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST)> 2.5 X institutional upper limit of normal (IULN). Total bilirubin > 1.5 X IULN (unless Gilbert syndrome has been diagnosed)
* Inadequate renal function (serum Cr >3 UNL or ClCr <45 ml/min)
* Patients receiving concurrent treatment with other experimental drugs or anti-cancer therapy
* Patients with uncontrolled concurrent disease:

Known pleural effusion at baseline Clinically-significant gastrointestinal disease or surgery that would compromise absorption of study drug (eg, uncontrolled nausea or malabsorption syndrome) Clinically-significant known coagulation or platelet function disorder (not related to thrombocytopenia), eg, von Willebrand's disease Other active malignancy requiring concurrent intervention

Uncontrolled or significant cardiovascular disease, including any of the following:

Myocardial infarction within 6 months of enrolment date Uncontrolled angina or congestive heart failure within 3 months of enrolment date Left ventricular ejection fraction (LVEF) < 40% Significant cardiac conduction abnormality, including history of clinically-significant ventricular arrhythmia (such as ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes), history of third degree heart block or diagnosed congenital long QT syndrome, and/or prolonged QTc/f interval > 450 msec on baseline ECG.

* Patients with active or uncontrolled infections or with serious illnesses or medical conditions that would not permit the patient to be managed according to the protocol.
* Patients unable or unwilling to give written, informed consent prior to study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Asses the efficacy | 1 year
  To assess the efficacy of dasatinib in terms of major molecular response rate at 6 months in patients with CP-CML who have achieved complete cytogenetic response without major molecular response after at least 18 months on Imatinib 400/600

SECONDARY OUTCOMES:
Asses the efficacy | 1 year
  To assess the efficacy of dasatinib in terms of depth and kinetics of molecular response
Assess the relationship of dasatinib with the appearance of large granular lymphocytes | 6 months
  To assess the relationship of dasatinib with the appearance of large granular lymphocytes and assess the relationship of LGL with efficacy and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Steegmann Juan Luis, Dr, Study Chair — PETHEMA Foundation; García Valentín, Dr, Study Chair — PETHEMA Foundation
Locations (15):
- Spain (15):
  - Hospital Txagorritxu, Vitoria-Gasteiz, Alava
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Institut Catalá d'Oncologia L'Hospitallet, Barcelona, Barcelona
  - Complejo Hospitalario de Toledo - Hospital Virgen de la Salud, Toledo, Castille-La Mancha
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital San Pedro de La Rioja, Logroño, La Rioja
  - Hospital de León, León, León
  - Hospital Universitario de la Princesa, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital POVISA, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Virgen del Rocío, Seville, Sevilla

REFERENCES:
- See also: Dynamic Solutions CRO — http://www.dynasolutions.com
- See also: Bristol Myers Squibb — http://www.bms.es